CLINICAL TRIAL: NCT06872060
Title: The Effects of Glucagon on Renal Regional Blood Flow in Humans Measured by Magnetic Resonance.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ali Asmar, Chief Physician, Associate Professor, PhD, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-24012271
Record Dates: First submitted 2025-02-21; First posted 2025-03-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Glucagon; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Glucagon (Experimental)
  Interventions: Drug: Glucagon; Drug: Glucagon+Exendin9-39; Drug: Sodium chloride
- Glucagon+Exendin9-39 (Experimental)
  Interventions: Drug: Glucagon; Drug: Glucagon+Exendin9-39; Drug: Sodium chloride
- Sodium chloride (Placebo comparator) (Placebo Comparator)
  Interventions: Drug: Glucagon; Drug: Glucagon+Exendin9-39; Drug: Sodium chloride

INTERVENTIONS:
Drug: Glucagon — Glucagon infusion at 5 ng·kg-¹·min-¹ from 0-30 minutes and 10 ng·kg-¹·min-¹ from 30-60 minutes.
Drug: Glucagon+Exendin9-39 — Glucagon infusion at 5 ng·kg-¹·min-¹ from 0-30 minutes and 10 ng·kg-¹·min-¹ from 30-60 minutes, plus a GLP-1R antagonist, exendin 9-39 (900 pmol·kg-¹·min-¹), given intravenously from -30 to 60 minutes
Drug: Sodium chloride — Placebo (0.9% NaCl).

SUMMARY:
This study will investigating the effects of glucagon on renal blood flow in humans using MRI technology. Glucagon, a hormone produced by the pancreas, plays a key role in regulating blood sugar levels. It has been shown to affect renal function, including electrolyte balance and blood flow, especially in conditions like type 2 diabetes where abnormal glucagon levels are common. The study aims to understand how glucagon affects regional blood flow in the kidneys, specifically the cortex and medulla, and whether these effects are mediated by glucagon receptors.

The study will be conducted on 10 healthy male participants aged 20-60 years. It involves three test days where participants will receive either glucagon, glucagon with a GLP-1 receptor antagonist, or placebo. Blood flow, glomerular filtration rate, and other renal functions will be measured using MRI. The study seeks to clarify whether glucagon's effects on the kidneys are linked to changes in regional blood flow and to determine if these effects are mediated solely by glucagon receptors.

ELIGIBILITY:
Inclusion Criteria:

* Normal health confirmed through; Interview and Medical examination
* Normal values with respect to blood concentrations of fasting plasma glucose, fasting plasma total cholesterol, fasting triglycerides, HDL, LDL, creatinine, liver function tests, and electrolytes
* Informed consent

Exclusion Criteria:

* Immunosuppressive treatment in the previous 12 months
* Alcohol abuse
* Medical treatment with oral glucocorticoids, dipeptidyl peptidase-4 (DPP-4) inhibitors, or GLP-1 receptor agonists, which, in the opinion of the principal investigator, may interfere with glucose metabolism
* Use of lithium
* Medical treatment that affects insulin secretion or the renin-angiotensin-aldosterone system
* Liver disease (ALT > 2x normal value)
* Renal impairment (serum creatinine > 130 µM and/or albuminuria)
* Individuals with severe claustrophobia
* Individuals with MR-incompatible foreign bodies
* Individuals with hypertension

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Blood perfusion of the kidney | 7 measurements of 10 minutes each from the start of infusion (time 0) and up to one hour (time 60).
  we would like to measure blood perfusion of the kidneys over time

SECONDARY OUTCOMES:
Blood flow of the renal arteries | 7 measurements of 10 minutes each from the start of infusion (time 0) and up to one hour (time 60).
blood oxygen saturation of the kidneys | 7 measurements of 10 minutes each from the start of infusion (time 0) and up to one hour (time 60).

IPD SHARING:
Plan to Share IPD: No